CLINICAL TRIAL: NCT04266314
Title: Maternal Marijuana Use and Fetal and Infant Outcome
Status: Withdrawn | Type: Observational
Why Stopped: unable to enroll
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00190055
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cannabis Use Disorder; Pregnancy Related
Keywords: Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Maternal-fetal monitoring — Maternal-fetal monitoring evaluates fetal and maternal heart rate, maternal respirations, fetal movement, and maternal skin conductance (a way to monitor emotional response)
Other: NICU Network Neurobehavioral Scale — Evaluates neurobehavioral organization, neurological reflexes, motor development, and signs of stress and withdrawal of substance-exposed infants.

SUMMARY:
Marijuana and cannabis-containing products are growing in popularity and availability in the United States, and use during pregnancy has increased dramatically. The overarching aim of this proposal is to provide pilot data for a submission which will explore the impact of chronic maternal marijuana use (primary or secondary) on fetal functioning, maternal reflective functioning and infant birth and neurodevelopmental outcomes. Chronically marijuana using pregnant women in treatment at the Center for Addiction and Pregnancy will be enrolled and asked to provide information about participants' marijuana and other licit and illicit substance use and feelings about parenting and participants' infant and undergo fetal monitoring at 36 weeks gestation. The neonates will undergo neurobehavioral examination during the first and fourth weeks of life.

ELIGIBILITY:
Maternal Inclusion Criteria:

* Singleton pregnancy less than 36 weeks of gestation
* Marijuana as a primary or secondary drug of choice

Maternal Exclusion Criteria:

* Significant fetal anomaly
* Multiple gestation
* Delivery prior to 36 weeks gestation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronically marijuana using women enrolled at the Center for Addiction and Pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Prevalence of maternal cannabis use disorder | The first day of study enrollment and again at infant delivery
  Rates of Cannabis use disorder among pregnant women reporting primary or secondary (i.e. first or second drug of choice) cannabis use during pregnancy.
Fetal functioning as assessed by fetal heart rate | One day during 36th weeks of gestation
  Fetal heart rate in beats per minute will be measured.
Fetal functioning as assessed by fetal movement | One day during 36th weeks of gestation
  Fetal movement: number and length in msecs of bouts of fetal movement as determined by fetal actograph testing
Change in infant neurobehavioral functioning as assessed by the NICU Network Neurobehavioral Scale | One day during week 1 and week 4 of infant life
  Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale scores.
Change in Maternal reflective functioning as assessed by the Parental Reflective Functioning Questionnaire | At 36 weeks of gestation, postpartum week 1, postpartum week 4
  Responses that evaluate the mother's ability to reflect on and interpret her own behavior and that of her child in terms of mental states and intentions; this will be assessed using the Parental Reflective Functioning Questionnaire.
Infant weight at birth | At the time of delivery
  Birth weight in kilograms
Infant length at birth | At the time of delivery
  Infant length in centimeters
Infant head circumference at birth | At the time of delivery
  Infant head circumference in centimeters
Infant Apgar Score at 1 minute | At 1 minute after delivery
  Apgar Score after birth at one minute; scores range from 1-10 with higher scores signifying more optimal infant well being at birth.
Infant Apgar Score at 5 minutes | At 5 minutes after delivery
  Apgar Score after birth at five minutes; scores range from 1-10 with higher scores signifying more optimal infant well being at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pajulo M, Tolvanen M, Karlsson L, Halme-Chowdhury E, Ost C, Luyten P, Mayes L, Karlsson H. THE PRENATAL PARENTAL REFLECTIVE FUNCTIONING QUESTIONNAIRE: EXPLORING FACTOR STRUCTURE AND CONSTRUCT VALIDITY OF A NEW MEASURE IN THE FINN BRAIN BIRTH COHORT PILOT STUDY. Infant Ment Health J. 2015 Jul-Aug;36(4):399-414. doi: 10.1002/imhj.21523. Epub 2015 Jun 19. PMID 26096692
- [Background] Lester BM, Andreozzi-Fontaine L, Tronick E, Bigsby R. Assessment and evaluation of the high risk neonate: the NICU Network Neurobehavioral Scale. J Vis Exp. 2014 Aug 25;(90):3368. doi: 10.3791/3368. PMID 25177897